CLINICAL TRIAL: NCT06754748
Title: Investigating the Acute Impacts of Caffeinated Coffee, Decaffeinated Coffee, and Water on Body Composition Parameters Measured Via Bioelectrical Impedance Analysis
Brief Title: Acute Effects of Caffeinated and Decaffeinated Coffee on Bioelectrical Impedance Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Guleren Sabuncular, Principal Investigator, Marmara University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GS_1
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Body Composition Measurement
Keywords: Bioelectrical Impedance Analysis; Caffeine; Hydration; Body Composition
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeinated coffee (Experimental): Coffee made with 11 g caffeinated coffee and 200 ml water was given to participants. BIA measurement was done before and after coffee intake every 30 minutes up to 120 minutes.
  Interventions: Other: Caffeinated coffee
- Decaffeinated coffee (Experimental): Coffee made with 11 g decaffeinated coffee and 200 ml water was given to participants. BIA measurement was done before and after coffee intake every 30 minutes up to 120 minutes.
  Interventions: Other: Decaffeinated coffee
- Water (Experimental): 200 ml water was given to participants. BIA measurement was done before and after coffee intake every 30 minutes up to 120 minutes.
  Interventions: Other: Water

INTERVENTIONS:
Other: Caffeinated coffee — 11 g caffeinated coffee made with 200 ml water was given to participants.
  Arms: Caffeinated coffee
Other: Decaffeinated coffee — 11 g decaffeinated coffee made with 200 ml water was given to participants.
  Arms: Decaffeinated coffee
Other: Water — 200 ml water was given to participants.
  Arms: Water

SUMMARY:
This study investigates how caffeinated coffee, decaffeinated coffee, and water affect body composition, as measured by BIA. Participants were divided into three groups, consuming their respective beverages, with measurements taken over a 120-minute period. The study aimed to determine if caffeine or fluid intake is the primary driver of changes in body composition parameters.

DETAILED DESCRIPTION:
This study aims to address these gaps by examining how caffeinated coffee, decaffeinated coffee, and water influence BIA measurements at multiple intervals post-consumption (baseline, 30, 60, 90, and 120 minutes). By incorporating a controlled study design with separate water-only and caffeine-free groups, this methodology overcomes the limitations of previous studies that lacked comprehensive control conditions. By determining whether caffeine or fluid volume primarily drives changes in BIA parameters and identifying the timing of these effects, this research seeks to improve the understanding of external factors affecting BIA, providing valuable insights for accurate body composition assessments.

Participants were divided into three groups based on their average daily caffeine consumption: caffeinated coffee, decaffeinated coffee, and water.

To standardize caffeine and fluid intake, filter coffee was chosen for its consistency in caffeine content and fluid volume. Both caffeinated and decaffeinated Arabic coffee were prepared using 11 g of coffee per 200 ml of water. The coffee was weighed using a precision balance and brewed with a filter coffee machine to ensure uniform preparation.

Participants were instructed to adhere to the following restrictions prior to the analysis day: a 12-hour fast, avoidance of excessive fluids, abstinence from caffeine-containing beverages, no showering or sauna use, no alcohol consumption for 48 hours, and no heavy exercise for 4-12 hours before the measurement. These restrictions minimized potential confounding effects on hydration or metabolic state, ensuring reliable BIA measurements.

The first BIA measurements were taken before any beverage consumption. Subsequently, participants consumed 200 ml of caffeinated coffee, decaffeinated coffee, or water, depending on their group. BIA measurements were repeated at 30, 60, 90, and 120 minutes post-consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥18 years.
* BMI between 18.5 and 29.9 kg/m².
* Regular coffee consumers.
* Participants providing written informed consent.

Exclusion Criteria:

* Individuals on medication or hormone therapy within the last 6 months.
* Medical conditions affecting caffeine metabolism (e.g., allergies or intolerances).
* Chronic or acute diseases.
* Significant appetite or eating disturbances in the past 6 months.
* Participants menstruating on the day of analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Change in Body Fat Mass | Baseline, 30, 60, 90 and 120 minutes
  BIA measurements were recorded for the body fat mass (kg) at baseline, 30, 60, 90, and 120 minutes.
Change in body fat percentage | Baseline and 30, 60, 90, and 120 minutes.
  BIA measurements were recorded for the body fat percentage (%) at baseline, 30, 60, 90, and 120 minutes.
Change in fat-free mass | Baseline and 30, 60, 90, and 120 minutes.
  BIA measurements were recorded for the fat-free mass (kg) at baseline, 30, 60, 90, and 120 minutes.
Change in muscle mass | Baseline and 30, 60, 90, and 120 minutes.
  BIA measurements were recorded for the muscle mass (kg) at baseline, 30, 60, 90, and 120 minutes.
Change in total body water | Baseline and 30, 60, 90, and 120 minutes.
  BIA measurements were recorded for the total body water (kg) at baseline, 30, 60, 90, and 120 minutes.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline, 30, 60, 90 and 120 minutes
  Body weight (kg) was measured with BIA at baseline, 30, 60, 90 and 120 minutes and recorded.
Change in Body Mass Index | Baseline, 30, 60, 90 and 120 minutes
  Body mass index was calculated from weight and height and presented as kg/m² at baseline, 30, 60, 90 and 120 minutes and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Guleren Sabuncular, PhD, Study Director — Marmara University
Locations (1):
- Marmara University, Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No